CLINICAL TRIAL: NCT00520468
Title: Treatment of Myelodysplastic Syndrome (MDS) With Cytokine-Immunotherapy for Low-Risk MDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0253
Record Dates: First submitted 2007-08-23; First posted 2007-08-24 (Estimated); Results first posted 2011-04-14 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Myelodysplastic Syndrome
Keywords: Myelodysplastic Syndrome; MDS; Erythropoietin; Darbepoetin alfa; Aranesp; Erythropoiesis stimulating protein; G-CSF; Filgrastim; Neupogen; Prednisone; Cyclosporin A; Sandimmune; CYA; Cyclosporine
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Erythropoietin; Darbepoetin alfa; Cyclosporine; Granulocyte Colony-Stimulating Factor; Filgrastim; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cytokine-Immunotherapy (Experimental): Erythropoietin 40,000 units subcutaneously (SQ) weekly; G-CSF 300 mcg SQ twice a week; Prednisone 60 mg/Day for 7 days, taper over 1 month; Cyclosporin A 300 mg orally daily
  Interventions: Drug: Erythropoietin; Drug: Cyclosporin A; Drug: G-CSF; Drug: Prednisone

INTERVENTIONS:
Drug: Erythropoietin — 40,000 units injected under the skin (SQ) weekly
  Other Names: Darbepoetin alfa; Aranesp; Erythropoiesis stimulating protein
Drug: Cyclosporin A — 300 mg (tablets) by mouth daily for 6 months
  Other Names: CYA; Cyclosporine; Sandimmune
Drug: G-CSF — 300 mcg injected under the skin (SQ) two times per week
  Other Names: Filgrastim; Neupogen
Drug: Prednisone — 60 mg per day for 7 days, taper over 1 month

SUMMARY:
Objectives:

Primary: To evaluate the response rate of total cytokine-immunotherapy for low-risk myelodysplastic syndromes (MDS).

Secondary: To evaluate response duration, survival and side effects of the treatment.

DETAILED DESCRIPTION:
MDS is a disease that produces low blood counts and may cause anemia, infections, and/or bleeding. Erythropoietin and Granulocyte colony-stimulating factor (G-CSF or GCSF) are drugs that stimulate the production of red cells and white cells. Prednisone and cyclosporin are drugs that work against MDS by affecting your immune system.

Before you can start treatment on this study, you will have what are called "screening tests". These tests will help the doctor decide if you are eligible to take part in the study. You will have a complete medical history and physical exam. Routine blood tests (between 4-6 tablespoons) will be performed. You will have a bone marrow aspiration. To collect a bone marrow aspirate, an area of the hip or chest bone is numbed with anesthetic and a small amount of bone marrow is withdrawn through a large needle. Women who are able to have children must have a negative blood or urine pregnancy test.

If you are found to be eligible to take part in this study, you will receive erythropoietin as an injection under the skin once a week and G-CSF as an injection under the skin 1-2 times a week for as long as you respond well to treatment. You will take prednisone by mouth every day for a month and cyclosporin tablets by mouth every day for 6 months.

During this study, you will need to visit your doctor for a physical exam and measurement of your vital signs. The frequency of doctor visits will vary depending on your physical condition, but will be required at least once every 3 months.

Blood tests (about 2 teaspoons) will be done about every 1-2 weeks during the first 12 weeks of treatment, then every 2 to 4 weeks for the remainder of the study. The blood samples will be collected for routine lab tests. Periodic (every 3 to 6 months) bone marrow samples will also be taken to check cells related to the disease before, during, and after completion of this study.

You will be taken off study if the disease gets worse or intolerable side effects occur.

This is an investigational study. All drugs are FDA approved and commercially available. Up to 60 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with MDS and </= 10% blasts or International Prognostic Scoring System (IPSS) low or intermediate 1. No prior intensive chemotherapy or high-dose ara-C (>/= 1g/m2). Prior cytokines, biologic therapies, targeted therapies, or single agent chemotherapy allowed. Procrit, G-CSF are allowed before therapy. Patients with blasts < 5% must have an indication for therapy, such as transfusion needs, symptomatic anemia or Hb < 11g/dl, platelets < 100 x 10 9/L, or granulocytes < 10 9/L.
2. Performance 0-2 (Eastern Cooperative Oncology Group (ECOG)). Adequate liver function (bilirubin of < 2mg/dl) and renal function (creatinine < 2mg/dl). Adequate cardiac functions (New York Heart Association (NYHA) cardiac III-IV excluded)
3. Signed informed consent

Exclusion Criteria:

1. Nursing and pregnant females are excluded. Women of childbearing potential should practice effective methods of contraception. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
2. Patients with active and uncontrolled infections.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2004-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gautam Borthakur, MBBS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Anderson Cancer Center's Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period 6/15/04 - 6/1/09; all patients were registered at The University of Texas M.D. Anderson Cancer Center.
Pre-assignment Details: Of fifteen patients enrolled, fourteen patients registered were evaluable and one patient taken off study never having received study drug.
Groups:
- Cytokine-Immunotherapy: Erythropoietin 40,000 units subcutaneously (SQ) weekly; G-CSF 300 mcg SQ twice per week; Prednisone 60 mg/Day for 7 days, taper over 1 month; Cyclosporin A 300 mg orally daily
Period: Overall Study
Arm/Group | Cytokine-Immunotherapy
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cytokine-Immunotherapy
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 8
Age Continuous [Mean (Full Range); unit: Years] | 65 [47 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Response
Description: Periodic bone marrow samples (every 3-6 months) to check cells related to disease before/during/after study. Response classifications categorized by the International Working Group Response Criteria for Myelodysplastic Syndrome (MDS) as: Complete Remission, Partial Response, Hematologic Improvement or No Response.
Time Frame: Response evaluation within first 3 months from start of therapy, then every 3 to 6 months
Population: All treated patients on study included in analysis.
Measure: Number; unit: participants
Arm/Group | Cytokine-Immunotherapy
Number analyzed (Participants) | 14
participants
  Complete Remission | 2
  Partial Response | 2
  Hematologic Improvement | 4
  No Response | 6

ADVERSE EVENTS:
Time Frame: 2 years 2 months
Arm/Group | Cytokine-Immunotherapy
Serious Adverse Events (participants affected / at risk) | 11/14
Other Adverse Events (participants affected / at risk) | 11/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cytokine-Immunotherapy (N=14)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Pain (General disorders) | 1 (1)
hemorrhage (Vascular disorders) | 3 (3)
Elevated creatinine (Blood and lymphatic system disorders) | 2 (2)
Chest Pain (General disorders) | 4 (4)
Fever (General disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Dizziness (General disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cytokine-Immunotherapy (N=14)
Hypertension (Cardiac disorders) | 3 (3)
elevated creatinine (Blood and lymphatic system disorders) | 3 (3)
Pain (General disorders) | 5 (6)
Hypomagnesemia (Blood and lymphatic system disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Insomnia (Nervous system disorders) | 1 (1)
Puritis (Skin and subcutaneous tissue disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Hyperbilirubinemia (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No